CLINICAL TRIAL: NCT05091567
Title: A Phase III, Randomized, Open-Label, Multicenter Study of Lurbinectedin in Combination With Atezolizumab Compared With Atezolizumab as Maintenance Therapy in Participants With Extensive-Stage Small-Cell Lung Cancer (ES-SCLC) Following First-Line Induction Therapy With Carboplatin, Etoposide and Atezolizumab
Brief Title: A Phase III, Open-Label Study of Maintenance Lurbinectedin in Combination With Atezolizumab Compared With Atezolizumab in Participants With Extensive-Stage Small-Cell Lung Cancer
Acronym: IMforte
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO43104; 2023-503868-16-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Small-Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; PM 01183; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Atezolizumab+Lurbinectedin (Experimental): Induction phase: participants will receive standard of care atezolizumab on Day 1 of each 21-day cycle in combination with carboplatin on Day 1 and etoposide on Days 1, 2, and 3 of each 21-day cycle for 4 cycles.
  Maintenance phase: participants will receive atezolizumab on Day 1 of each 21-day cycle in combination with lurbinectedin on Day 1 of each 21-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Lurbinectedin; Drug: Carboplatin; Drug: Etoposide
- Arm B: Atezolizumab (Active Comparator): Induction phase: participants will receive standard of care atezolizumab on Day 1 of each 21-day cycle in combination with carboplatin on Day 1 and etoposide on Days 1, 2, and 3 of each 21-day cycle for 4 cycles.
  Maintenance phase: participants will receive atezolizumab on Day 1 of each 21-day cycle.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered intravenously at a fixed dose of 1200 mg on Day 1 of each 21-day cycle for 4 cycles in the induction phase. Atezolizumab will be administered intravenously at a fixed dose of 1200 mg on Day 1 of each 21-day cycle in the maintenance phase.
  Other Names: Tecentriq, RO5541267
Drug: Lurbinectedin — Lurbinectedin 3.2 mg/m² will be administered intravenously on Day 1 of each 21-day cycle in the maintenance phase.
  Other Names: PM01183/JZP712
  Arms: Arm A: Atezolizumab+Lurbinectedin
Drug: Carboplatin — Carboplatin will be administered according to the standard of care treatment for 4 cycles in the induction phase.
Drug: Etoposide — Etoposide will be administered according to the standard of care treatment for 4 cycles in the induction phase.

SUMMARY:
Study GO43104 is a Phase III, randomized, open-label, multicenter study of lurbinectedin in combination with atezolizumab compared with atezolizumab alone administered as maintenance therapy in participants with extensive-stage small-cell lung cancer (ES-SCLC) after first-line induction therapy with carboplatin, etoposide, and atezolizumab. The study consists of 2 phases: an induction phase and a maintenance phase. Participants need to have an ongoing response or stable disease per the Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 criteria after completion of 4 cycles of carboplatin, etoposide, and atezolizumab induction treatment in order to be considered for eligibility screening for the maintenance phase. Eligible participants will be randomized in a 1:1 ratio to receive either lurbinectedin plus atezolizumab or atezolizumab in the maintenance phase.

ELIGIBILITY:
Inclusion Criteria for the Induction Phase:

* ECOG PS of 0 or 1
* No prior systemic therapy for ES-SCLC
* Treatment-free for at least 6 months since last chemo/radiotherapy, among those treated (with curative intent) with prior chemo/radiotherapy for limited-stage SCLC
* Histologically or cytologically confirmed ES-SCLC
* Adequate hematologic and end-organ function to receive 4 cycles of induction treatment with carboplatin, etoposide and atezolizumab
* Measurable disease, as defined by RECIST v1.1
* Negative HIV test and no evidence of active Hepatitis B or Hepatitis C at screening

Exclusion Criteria for the Induction Phase:

* Presence or history of CNS metastases
* Active or history of autoimmune disease or deficiency
* History of malignancies other than SCLC within 5 years prior to enrollment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, or lurbinectedin or trabectedin
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Treatment with investigational therapy within 28 days prior to enrollment

Inclusion Criteria for the Maintenance Phase:

* ECOG PS of 0 or 1
* Ongoing response or stable disease per RECIST 1.1 after 4 cycles of induction therapy
* Toxicities attributed to prior induction anti-cancer therapy or PCI resolved to Grade <=1
* Adequate hematologic and end-organ function

Exclusion Criteria for the Maintenance Phase:

* Presence or history of CNS metastases
* Receiving consolidative chest radiation
* Severe infection within 2 weeks prior to randomization into the maintenance
* Treatment with therapeutic oral or IV antibiotics at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2026-08-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (94):
- United States (14):
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Marietta, Georgia
  - Illinois Cancer Care, Peoria, Illinois
  - New England Cancer Specialists, Scarborough, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Mercy Research - St. Louis, St Louis, Missouri
  - Clinical Research Alliance, Westbury, New York
  - The Mark H. Zangmeister Ctr, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center, Charleston, South Carolina
  - Greco-Hainesworth Centers for Research, Chattanooga, Tennessee
  - West Clinic, Germantown, Tennessee
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
- Belgium (6):
  - Institut Jules Bordet, Anderlecht
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - UZ Leuven Gasthuisberg, Leuven
  - AZ St Maarten Campus Leopoldstr, Mechelen
  - CHU UCL Mont-Godinne, Mont-godinne
  - Vitaz, Sint-Niklaas
- Germany (11):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - KEM/Evang. Kliniken Essen Mitte gGmbH, Essen
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg GmbH, Georgsmarienhütte
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Asklepios Klinik Gauting, München-Gauting
- Greece (6):
  - Sotiria Thoracic Diseases Hospital of Athens, Athens
  - Errikos Dynan Hospital, Athens
  - University Hospital of Larissa, Larissa
  - Euromedical General Clinic of Thessaloniki, Thessaloniki
  - Ag. Loukas Hospital, Thessaloniki
  - Diavalkaniko Hospital, Thessaloniki
- Hungary (4):
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Pécsi Tudományegyetem, Pécs
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rend.Int., Szolnok
  - Tudogyogyintezet Torokbalint, Törökbálint
- Italy (5):
  - AUSL della Romagna, Ravenna, Emilia-Romagna
  - ASL 3 Genovese, Genoa, Liguria
  - Irccs Istituto Europeo di Oncologia (IEO), Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Ospedale Niguarda Ca' Granda), Milan, Lombardy
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette Di Ancona, The Marches
- Mexico (2):
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Morelia
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Krakowski Szpital Specjalistyczny im sw. Jana Paw?a II, Krakow
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan
  - Centrum Onkologii Instytut im.Marii Sklodowskiej-Curie, Warsaw
- South Korea (8):
  - Chungbuk National University Hospital, Cheongju-si
  - Chilgok Kyungpook National University Medical Center, Daegu
  - Samsung Changwon Hospital, Gyeongsangnam-do
  - Gyeongsang National University Hospital, Gyeongsangnam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (7):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (4):
  - E-DA Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (15):
  - Adana Baskent University Hospital, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Liv Hospital Ankara, Ankara
  - Ankara City Hospital, Ankara
  - Uludag Uni Hospital, Bursa
  - Pamukkale University School Of Medicine, Denizli
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Ba?c?lar Medipol Mega Üniversite Hastanesi, Istanbul
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital, Istanbul
  - Ac?badem Altunizade Hastanesi, Istanbul
  - Izmir Medical Point Hospital, Izmir
  - Kocaeli University Faculty of Medicine, İzmit
  - Goztepe Prof.Dr. Suleyman Yalcin City Hospital, Kadiköy
  - Medikal Park Samsun, Samsun
  - TC Necmettin Erbakan University Meram Medical Faculty Hospital, Selçuklu
- United Kingdom (6):
  - Blackpool Victoria Hospital, Blackpool
  - Christie NHS Foundation Trust, GB Manchester
  - Castle Hill Hospital, Hull
  - St James University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Paz-Ares L, Borghaei H, Liu SV, Peters S, Herbst RS, Stencel K, Majem M, Sendur MAN, Czyzewicz G, Caro RB, Lee KH, Johnson ML, Karadurmus N, Grohe C, Baka S, Csoszi T, Ahn JS, Califano R, Yang TY, Kemal Y, Ballinger M, Cuchelkar V, Graupner V, Lin YC, Chakrabarti D, Bhatt K, Cai G, Iannone R, Reck M; IMforte investigators. Efficacy and safety of first-line maintenance therapy with lurbinectedin plus atezolizumab in extensive-stage small-cell lung cancer (IMforte): a randomised, multicentre, open-label, phase 3 trial. Lancet. 2025 Jun 14;405(10495):2129-2143. doi: 10.1016/S0140-6736(25)01011-6. Epub 2025 Jun 2. PMID 40473449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 660 participants with ES SCLC took part in the study across 96 investigative sites in 13 countries.
Pre-assignment Details: The study consists of 2 phases, an enrollment phase (induction phase), where participants received standard of care treatment with carboplatin, etoposide and atezolizumab, and a randomized phase (maintenance phase), where participants were randomized in 1:1 ratio to receive either atezolizumab + lurbinectedin or atezolizumab. The study is ongoing.
Groups:
- Atezolizumab + Carboplatin + Etoposide: Participants received atezolizumab, 1200 milligrams (mg), every 3 weeks (Q3W) as intravenous (IV) infusion on Day 1 of each 21-day cycle in combination with carboplatin on Day 1 and etoposide, in accordance with local standard of care, on Days 1, 2, and 3 of each cycle for up to 4 cycles.
- Atezolizumab: Participants received atezolizumab, 1200 mg, Q3W as IV infusion on Day 1 of each 21-day cycle until unacceptable toxicity or disease progression (PD) whichever occurred first.
- Atezolizumab+ Lurbinectedin: Participants received atezolizumab, 1200 mg, Q3W as IV infusion and lurbinectedin, 3.2 milligrams per square meter (mg/m^2), Q3W as IV infusion on Day 1 of each 21-day cycle until unacceptable toxicity or PD whichever occurred first.
Period: Enrollment Phase
Arm/Group | Atezolizumab + Carboplatin + Etoposide | Atezolizumab | Atezolizumab+ Lurbinectedin
Started | 660 | 0 | 0
Enrolled Safety Analysis Set (SAS) (Enrolled SAS included all enrolled participants who received at least 1 dose of treatment, regardless of whether/not, they were randomized.) | 653 | 0 | 0
Completed | 571 | 0 | 0
Not Completed | 89 | 0 | 0
Not completed — Death | 37 | 0 | 0
Not completed — Adverse Event | 21 | 0 | 0
Not completed — Progressive Disease | 10 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0
Not completed — Symptomatic Deterioration | 7 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Reason not Specified | 1 | 0 | 0
Period: Randomized Phase
Arm/Group | Atezolizumab + Carboplatin + Etoposide | Atezolizumab | Atezolizumab+ Lurbinectedin
Started | 0 | 241 | 242
SAS (SAS included all participants who were randomized & received at least 1 dose of atezolizumab/lurbinectedin.) | 0 | 240 | 242
Completed | 0 | 0 | 0
Not Completed | 0 | 241 | 242
Not completed — Death | 0 | 135 | 112
Not completed — Progressive Disease | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Ongoing in Study | 0 | 102 | 126

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants randomized into the randomized phase, regardless of whether or not the assigned study treatment was received. Analysis was performed on the randomized treatment arms.
Groups:
- Atezolizumab: Participants received atezolizumab, 1200 mg, Q3W as IV infusion on Day 1 of each 21-day cycle until unacceptable toxicity or PD whichever occurred first.
- Atezolizumab+ Lurbinectedin: Participants received atezolizumab, 1200 mg, Q3W, as IV infusion and lurbinectedin, 3.2 mg/m^2, Q3W, as IV infusion on Day 1 of each 21-day cycle until unacceptable toxicity or PD whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin | Total
Number analyzed (Participants) | 241 | 242 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (8.0) | 65.1 (7.6) | 65.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 91 | 181
  Male | 151 | 151 | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 32
  Not Hispanic or Latino | 210 | 206 | 416
  Unknown or Not Reported | 15 | 20 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 31 | 31 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 199 | 195 | 394
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Randomized Phase: Independent Review Facility (IRF) - Assessed Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the date of first documented PD as determined by the IRF according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) or death, whichever occurs first. PD was defined as appearance of a new lesion(s), unequivocal progression in non-target lesion(s) or at least a 20% increase in the sum of diameters (SOD) of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimetres (mm).
Time Frame: Up to 26 months
Population: FAS included all participants randomized into the randomized phase, regardless of whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 241 | 242
months | 2.14 (1.64) [1.64 to 2.73] | 5.36 (4.24) [4.24 to 5.75]
Statistical Analysis 1: Comparison: Atezolizumab vs Atezolizumab+ Lurbinectedin; Stratified Analysis: The stratification factors were Eastern Cooperative Oncology Group performance status (ECOG PS) at randomization (0 vs. 1); Lactate Dehydrogenase (LDH) at randomization (<=upper limit of normal (ULN) vs >ULN) via local laboratory test; Presence of liver metastases at enrollment (yes vs. no); Prior receipt of prophylactic cranial irradiation (PCI) (yes vs. no); Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.43 to 0.67]

2. Primary Outcome: Randomized Phase: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death from any cause.
Time Frame: Up to 26 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Atezolizumab+ Lurbinectedin: Participants received atezolizumab, 1200 mg, Q3W as IV infusion and lurbinectedin, 3.2 mg/m^2, Q3W as IV infusion on Day 1 of each 21-day cycle until unacceptable toxicity or PD whichever occurred first.
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 241 | 242
months | 10.64 (9.49) [9.49 to 12.16] | 13.24 (11.89) [11.89 to 16.36]
Statistical Analysis 1: Comparison: Atezolizumab vs Atezolizumab+ Lurbinectedin; Stratified Analysis: The stratification factors were ECOG PS at randomization (0 vs. 1); LDH at randomization (<=ULN vs >ULN) via local laboratory test; Presence of liver metastases at enrollment (yes vs. no); Prior receipt of PCI (yes vs. no); Test type: Superiority; p = 0.0174, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.57 to 0.95]

3. Secondary Outcome: Randomized Phase: Investigator-assessed PFS
Description: PFS was defined as the time from randomization to the date of first documented PD as assessed by investigator according to RECIST v1.1 or death, whichever occurs first. PD was defined as appearance of a new lesion(s), unequivocal progression in non-target lesion(s) or at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 26 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 241 | 242
months | 2.73 (2.53) [2.53 to 2.83] | 5.36 (4.30) [4.30 to 6.57]
Statistical Analysis 1: Comparison: Atezolizumab vs Atezolizumab+ Lurbinectedin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.45 to 0.68]

4. Secondary Outcome: Randomized Phase: Confirmed Objective Response Rate (ORR) as Determined by the IRF
Description: ORR was defined as the percentage of participants with an objective tumor response of complete response (CR) or partial response (PR) as determined by the IRF using RECIST v.1.1. CR was defined as the disappearance of all target and non-target lesions or any pathological lymph nodes (whether target or non-target) have a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD. Percentages have been rounded off.
Time Frame: Up to 26 months
Population: FAS included all participants randomized into the randomized phase, regardless of whether or not the assigned study treatment was received. Overall number analyzed is the number of participants with measurable disease at baseline, as assessed by IRF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 182 | 175
percentage of participants | 10.4 (6.40) [6.40 to 15.82] | 19.4 (13.85) [13.85 to 26.08]
Statistical Analysis 1: Comparison: Atezolizumab vs Atezolizumab+ Lurbinectedin; Stratified Analysis: The stratification factors were ECOGPS at randomization (0 vs. 1);LDH at randomization (<=ULN vs >ULN) via local laboratory test; Presence of liver metastases at enrollment (yes vs. no); Prior receipt of PCI (yes vs. no); Test type: Superiority; Difference in Overall Response Rates = 8.99, 95% CI 2-sided [1.07 to 16.90]

5. Secondary Outcome: Randomized Phase: Confirmed ORR as Determined by the Investigator
Description: ORR was defined as the percentage of participants with an objective tumor response of CR or PR as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) have a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD.
Time Frame: Up to 26 months
Population: FAS included all participants randomized into the randomized phase, regardless of whether or not the assigned study treatment was received. Overall number analyzed is the number of participants with measurable disease at baseline, as assessed by investigator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 205 | 205
percentage of participants | 13.2 (8.86) [8.86 to 18.58] | 17.1 (12.19) [12.19 to 22.94]
Statistical Analysis 1: Comparison: Atezolizumab vs Atezolizumab+ Lurbinectedin; Stratified Analysis: The stratification factors were ECOGPS at randomization (0 vs. 1);LDH at randomization (<=ULNvs >ULN) via local laboratory test; Presence of liver metastases at enrollment (yes vs. no); Prior receipt of PCI (yes vs. no); Test type: Superiority; Difference in Overall Response Rates = 3.90, 95% CI 2-sided [-3.51 to 11.32]

6. Secondary Outcome: Randomized Phase: Duration of Response (DOR) as Determined by the IRF
Description: DOR was calculated for participants who had a best confirmed OR of CR/PR. DOR= time from first occurrence of a documented OR until the time of documented PD as determined by IRF assessment using RECIST v1.1 or death from any cause, whichever occurs first. CR=disappearance of all target and non-target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR= at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD was defined as appearance of a new lesion(s), unequivocal progression in non-target lesion(s) or at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 26 months
Population: FAS included all participants randomized into the randomized phase, regardless of whether or not the assigned study treatment was received. Overall number analyzed is the number of participants with response, per IRF.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 19 | 34
months | 5.62 [4.17 to NA] — Upper limit of 95 %Cl was not estimable due to insufficient number of participants with events. | 9.00 [5.52 to NA] — Upper limit of 95 %Cl was not estimable due to insufficient number of participants with events.

7. Secondary Outcome: Randomized Phase: DOR as Determined by the Investigator
Description: DOR was calculated for participants who had a best confirmed OR of CR/PR. DOR= time from first occurrence of a documented OR until the time of documented PD as determined by investigator using RECIST v1.1 or death from any cause, whichever occurs first. CR=disappearance of all target and non-target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR= at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD was defined as appearance of a new lesion(s), unequivocal progression in non-target lesion(s) or at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 26 months
Population: FAS included all participants randomized into the randomized phase, regardless of whether or not the assigned study treatment was received. Overall number analyzed is the number of participants with response, per investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 27 | 35
months | 11.93 [8.38 to NA] — Upper limit of 95 %Cl was not estimable due to insufficient number of participants with events. | 5.75 [4.17 to 11.10]

8. Secondary Outcome: Randomized Phase: Percentage of Participants With PFS as Determined by the IRF at 6 Months and 12 Months
Description: PFS rate at 6 months and 12 months was defined as the percentage of participants who had not experienced PD as determined by the IRF according to RECIST v1.1 or death from any cause at 6 months and 12 months after randomization. PD was defined as appearance of a new lesion(s), unequivocal progression in non-target lesion(s) or at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Percentages have been rounded off.
Time Frame: Months 6 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 241 | 242
percentage of participants
  6 Months | 18.66 (13.45) [13.45 to 23.87] | 41.22 (34.58) [34.58 to 47.86]
  12 Months | 12.03 (7.27) [7.27 to 16.80] | 20.54 (14.37) [14.37 to 26.72]
Statistical Analysis 1: Comparison: Atezolizumab vs Atezolizumab+ Lurbinectedin; Test type: Superiority; Difference in Event Free Rate = 22.56, 95% CI 2-sided [14.12 to 31.00]
Statistical Analysis 2: Comparison: Atezolizumab vs Atezolizumab+ Lurbinectedin; Test type: Superiority; Difference in Event Free Rate = 8.51, 95% CI 2-sided [0.72 to 16.31]

9. Secondary Outcome: Randomized Phase: Percentage of Participants With PFS Determined by Investigator at 6 Months and 12 Months
Description: PFS rate at 6 months and 12 months was defined as the percentage of participants who had not experienced PD as determined by the investigator according to RECIST v1.1 or death from any cause at 6 months and 12 months after randomization. PD was defined as appearance of a new lesion(s), unequivocal progression in non-target lesion(s) or at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Percentages have been rounded off.
Time Frame: Months 6 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 241 | 242
percentage of participants
  6 Months | 22.56 (17.12) [17.12 to 28.00] | 46.21 (39.60) [39.60 to 52.81]
  12 Months | 12.80 (8.07) [8.07 to 17.52] | 20.32 (14.33) [14.33 to 26.32]
Statistical Analysis 1: Comparison: Atezolizumab vs Atezolizumab+ Lurbinectedin; Test type: Superiority; Difference in Event Free Rate = 23.65, 95% CI 2-sided [15.09 to 32.20]
Statistical Analysis 2: Comparison: Atezolizumab vs Atezolizumab+ Lurbinectedin; Test type: Superiority; Difference in Event Free Rate = 7.53, 95% CI 2-sided [-0.11 to 15.16]

10. Secondary Outcome: Randomized Phase: Percentage of Participants With OS at 12 Months and 24 Months
Description: OS rate at 12 months and 24 months was defined as the percentage of participants who had not experienced death from any cause at 12 months and 24 months after randomization. Percentages have been rounded off.
Time Frame: Months 12 and 24
Reporting Status: Not Posted

11. Secondary Outcome: Randomized Phase: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI)
Description: An AE =any unfavorable & unintended sign (including abnormal laboratory values/abnormal clinical test results), symptoms/disease temporally associated with the use of a pharmaceutical product, whether considered related to the pharmaceutical product. SAE=any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above. AESI= drug induced liver injury, suspected transmission of infectious agent via study treatment, hepatitis, systemic lupus erythematosus, hypersensitivity, etc. AESIs may include events not specified in the protocol.
Time Frame: Up to 26 months
Population: Saftey analysis set (SAS)=all participants who were randomized & received at least 1 dose of atezolizumab/lurbinectedin.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 240 | 242
Participants
  AEs | 194 | 235
  SAEs | 41 | 75
  AESIs for Atezolizumab | 54 | 76
  AESIs for Lurbinectedin | 62 | 93

12. Secondary Outcome: Randomized Phase: Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: For determining post-baseline incidence, participants were considered to be ADA-positive if they were ADA-negative or had missing data at baseline but developed at least one positive post-baseline ADA result during the randomized phase, or if they were ADA-positive at baseline and the titer of 1 or more post-baseline samples was at least 0.60 titer units (t.u.) greater than the baseline titer result.
Time Frame: Up to 26 months
Population: ADA-evaluable population was defined as participants with at least one post-dose evaluable ADA sample (collected in the randomized phase).
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 239 | 242
Participants | 20 | 19

13. Secondary Outcome: Randomized Phase: Time to Confirmed Deterioration (TTCD) in Physical Functioning (PF) and Global Health Status (GHS) as Measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQC30)
Description: EORTC QLQ-C30=30 questions assessing 5 aspects of participant functioning(physical,emotional,role,cognitive &social),3 symptom scales,GHS/QoL & 6 single items.PF scale=5 questions about participants PF & daily activities(strenuous activities,long walks,short walks,bed/chair rest & needing help with eating,dressing,washing themselves/using the toilet).PF scale scored on 4-point scale(1=Not at All-4=Very Much).GHS/QoL scored on 7-point scale(1=Very Poor- 7=Excellent).Scores were linearly transformed to a range of 0-100,higher scores=higher response level & better QoL.TTCD for PF & GHS/QoL=time from the date of randomization until first confirmed clinically meaningful deterioration,which is decrease from baseline in PF/GHS score that must be held for at least 2 consecutive assessments/initial decrease above baseline followed by death attributable to cancer progression within 6 weeks of the last deteriorated assessment.Score change≥10-point change in subscale score,considered meaningful.
Time Frame: Up to 26 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Atezolizumab+ Lurbinectedin
Number analyzed (Participants) | 241 | 242
months
  TTCD for PF | NA [NA to NA] — Percentage and 95 %Cl was not estimable due to insufficient number of participants with events. | 15.9 [11.0 to NA] — Upper limit of 95 %Cl was not estimable due to insufficient number of participants with events.
  TTCD for GHS/QoL | 12.9 [11.6 to NA] — Upper limit of 95 %Cl was not estimable due to insufficient number of participants with events. | 10.8 [7.6 to NA] — Upper limit of 95 %Cl was not estimable due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Enrollment Phase: Up to 6 months Randomization Phase: up to 26 months Study is ongoing & data up to primary clinical cut-off date is reported. Final data to be reported 1 year after study completion.
Description: All-Cause Mortality was assessed on all participants enrolled in the study.
  AE & SAE:Enrolled SAS=all enrolled participants who received at least 1 dose of treatment, regardless of whether/not, they were randomized. SAS=all participants who were randomized & received at least 1 dose of atezolizumab/lurbinectedin.
Groups:
- Atezolizumab + Carboplatin + Etoposide: Participants received atezolizumab, 1200 mg, Q3W as IV infusion on Day 1 of each 21-day cycle in combination with carboplatin on Day 1 and etoposide, in accordance with local standard of care, on Days 1, 2, and 3 of each cycle for up to 4 cycles.
Arm/Group | Atezolizumab + Carboplatin + Etoposide | Atezolizumab | Atezolizumab+ Lurbinectedin
All-Cause Mortality (participants affected / at risk) | 54/660 | 135/241 | 113/242
Serious Adverse Events (participants affected / at risk) | 181/653 | 41/240 | 75/242
Other Adverse Events (participants affected / at risk) | 526/653 | 127/240 | 213/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Carboplatin + Etoposide (N=653) | Atezolizumab (N=240) | Atezolizumab+ Lurbinectedin (N=242)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 22 (24) | 6 (6) | 6 (6)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular access site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Bacteroides infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 11 (11) | 1 (1) | 1 (1)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (13) | 3 (3) | 2 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (3)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (5) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 4 (4) | 0 (0) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 4 (4) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 3 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 3 (3)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1)
Administration site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 3 (3) | 0 (0) | 0 (0)
Adhesion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Perinephric collection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 25 (31) | 0 (0) | 2 (2)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 22 (23) | 0 (0) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric symptom (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Carboplatin + Etoposide (N=653) | Atezolizumab (N=240) | Atezolizumab+ Lurbinectedin (N=242)
Alopecia (Skin and subcutaneous tissue disorders) | 108 (110) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (34) | 17 (20) | 18 (20)
Hypothyroidism (Endocrine disorders) | 15 (15) | 17 (22) | 17 (18)
Asthenia (General disorders) | 68 (81) | 15 (19) | 31 (47)
Fatigue (General disorders) | 76 (88) | 19 (21) | 48 (59)
Hypomagnesaemia (Metabolism and nutrition disorders) | 48 (60) | 5 (5) | 12 (18)
Hyponatraemia (Metabolism and nutrition disorders) | 34 (42) | 11 (14) | 11 (19)
Decreased appetite (Metabolism and nutrition disorders) | 67 (69) | 16 (18) | 41 (51)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 (46) | 15 (15) | 19 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (30) | 16 (16) | 23 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 59 (84) | 4 (4) | 30 (53)
Anaemia (Blood and lymphatic system disorders) | 268 (319) | 16 (16) | 75 (116)
Neutropenia (Blood and lymphatic system disorders) | 110 (162) | 4 (6) | 26 (42)
Vomiting (Gastrointestinal disorders) | 35 (40) | 6 (6) | 33 (49)
Diarrhoea (Gastrointestinal disorders) | 55 (62) | 18 (21) | 34 (41)
Nausea (Gastrointestinal disorders) | 114 (138) | 9 (9) | 86 (151)
Constipation (Gastrointestinal disorders) | 90 (103) | 13 (13) | 27 (32)
Dizziness (Nervous system disorders) | 17 (21) | 5 (5) | 16 (20)
Headache (Nervous system disorders) | 14 (14) | 6 (6) | 15 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (21) | 12 (13) | 19 (21)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 16 (18)
Neutrophil count decreased (Investigations) | 102 (151) | 3 (3) | 31 (49)
Platelet count decreased (Investigations) | 49 (63) | 7 (7) | 35 (57)
Aspartate aminotransferase increased (Investigations) | 17 (20) | 11 (12) | 15 (18)
Blood creatinine increased (Investigations) | 18 (21) | 3 (3) | 13 (15)
White blood cell count decreased (Investigations) | 31 (46) | 5 (8) | 18 (32)
Alanine aminotransferase increased (Investigations) | 25 (28) | 9 (11) | 15 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT05091567/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT05091567/SAP_001.pdf